CLINICAL TRIAL: NCT05334264
Title: The Value of Prophylactic Cervical Cerclage Against Preterm Birth in Twin Pregnancies With History of Preterm Birth and Non-shortened Cervix: A Randomized Controlled Trial
Brief Title: Prophylactic Cervical Cerclage in Twin Pregnancies With Non-shortened Cervix
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hytham Atia, Associate professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ZU-IRB #8084/17-10-2021
Record Dates: First submitted 2021-12-11; First posted 2022-04-19 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Preterm Birth; Twin Pregnancy, Antepartum Condition or Complication; Cervical Cerclage
MeSH Terms: conditions — Premature Birth | interventions — Cerclage, Cervical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): cervical cerclage between 14 and 20 weeks will be done by one of the three authors. McDonald cervical cerclage.
  Interventions: Procedure: Cervical cerclage
- Group B (No Intervention): Routine antenatal care without cerclage

INTERVENTIONS:
Procedure: Cervical cerclage — McDonald cervical cerclage will be applied using Mersaline braided tape with double needle. Single stitch (4 bites) will be applied as close as possible to the level of internal os. The Knot will be put either anterior or posterior according to the surgeon desire.
  Arms: Group A

SUMMARY:
This randomized controlled trial is aimed to assess the protective value of prophylactic cervical cerclage against preterm birth in twin pregnancies with history of one or more preterm births without having cervical shortening in the current pregnancy.

DETAILED DESCRIPTION:
Multiple pregnancies are high-risk pregnancies and usually associated with an increased risk of neonatal morbidity and mortality, mainly due to preterm births. Preterm births occur in 50% of twin pregnancies and the mean gestational age for delivery is 35.3 weeks. Ten percent of all twin births take place before 32 weeks of gestation.1 Preterm births are responsible for more than 70% of all neonatal and infant deaths.2 Prematurity can have serious consequences for the child, such as hearing difficulties, vision impairment, learning disabilities, reduced IQ, and cerebral palsy. A cervical length of ≤25 mm in twin pregnancies is a good predictor of a spontaneous preterm birth when measured around 24 weeks of gestation.3,4 Numerous interventions have been attempted in order to prevent preterm births in twin gestations, but until now, no intervention has been effective. Use of cerclage in twin pregnancies is controversial. Some experts claim that placing a cervical cerclage could increase the risk of preterm births5, Fuchs and Senat6 concluded that cervical cerclage in asymptomatic twins did not reduce the risk of PTB. This conclusion came depending on small sample sized randomized trail done on less than 50 patients.7 Available meta-analytic data remained of limited value in view of the few and small clinical studies that were included.

Although the current meta-analyses indicate the lack of efficacy of cerclage in twin pregnancies, data from the US Standard Certificate of Live Birth indicated that roughly 10% of triplets and 1.3% of twins are still receiving cerclage.8 Some authors compared the efficacy of cerclage in twin pregnancies and singleton pregnancies and showed that women with twin pregnancies who received cerclage might show beneficial obstetric outcomes similar to those of women with singleton gestations.9,10 Such practice is still in need for further validation by well-structured and powered randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-50 years.
* Dichorionic twins.
* History of ≥1 preterm birth.
* Transvaginal sonographic cervical length is ≥25 mm at 14-20 weeks gestational age.
* Asymptomatic.

Exclusion Criteria:

* Triplets and quadruplets.
* Monochorionic twins.
* Threatened/ inevitable miscarriage
* Bulging membranes through the external os.
* Extremes of age.
* Major fetal anomalies.
* Known cases with uterine anomalies e.g. bicornuate uterus, uterus didelphis… etc.
* Fetal demise.
* Fetal reduction in the current pregnancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant ladies
Enrollment: 170 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
The incidence of preterm birth at ≤35+6, ≤33+6, and ≤31+6 weeks. | immediately after delivery for study cases through study completion, an average of 1 year
  Number of preterm deliveries stratified according to gestational age groups mentioned

SECONDARY OUTCOMES:
The incidence of miscarriage. | immediately after occurrence of miscarriage through study completion, an average of 1 year
  Number of missed, inevitable and complete miscarriage less than 20 weeks
Incidence of cervico-vaginal infection | once reported or confirmed during pregnancy through study completion, an average of 1 year
  Number of infections diagnosed by patient complaint, clinical examination and confirmed by culture and sensitivity
Incidences of bad Neonatal outcomes in both groups | during early neonatal follow up through study completion, an average of 1 year
  Number of of neonates with respiratory distress, IVH, necrotizing enterocolitis, sepsis, NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Amro El Nemr, Principal Investigator — Zagazig University; Mohamed Lashin, Principal Investigator — Zagazig University
Locations (1):
- Faculty of medicine, Zagazig University, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No